CLINICAL TRIAL: NCT03007537
Title: The Prevention of Erythropoietin on Cardiac Surgery-associated Acute Kidney Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSA-AKI2016
Record Dates: First submitted 2016-12-25; First posted 2017-01-02 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury; Cardiac Disease; Surgery
Keywords: Erythropoietin; Cardiac Surgery Associated-acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury; Heart Diseases | interventions — Erythropoietin; Sodium Chloride; Saline Solution; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): 0.9% sodium chloride 1ml, subcutaneous injection, once, applied 1day before cardiac surgery
  Interventions: Drug: 0.9% sodium chloride; Procedure: cardiac surgery
- Erythropoietin group (Experimental): 10000 IU erythropoietin, subcutaneous injection, once, applied 1day before cardiac surgery
  Interventions: Drug: Erythropoietin; Procedure: cardiac surgery

INTERVENTIONS:
Drug: Erythropoietin — 10000 IU erythropoietin, subcutaneous injection
  Other Names: EPO
  Arms: Erythropoietin group
Drug: 0.9% sodium chloride — 0.9% sodium chloride 1ml, subcutaneous injection
  Other Names: saline solution
  Arms: control group
Procedure: cardiac surgery — included valve, coronary artery bypass graft or surgery for congenital heart diseases
  Other Names: open-heart surgery

SUMMARY:
To testify the prevention of Erythropoietin on cardiac surgery associated-acute kidney injury, and trying to provide evidence for protecting the renal function and improving the prognosis for patients after cardiac surgery.

DETAILED DESCRIPTION:
Patients meet the inclusion criteria and agree to sign an informed consent will be randomly assigned into the control group or erythropoietin group.Interventions will be applied 1 day(24hrs) before the cardiac surgery. Blood and Urine samples will be collected after the surgery. By using the criterion given by KDIGO2012 and testing the biomarkers for acute kidney injury, we hope to find out if there is an association between erythropoietin administration and the occurence of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative hemoglobin<130g/L;
2. Surgery: valve, coronary artery bypass graft or surgery for congenital heart diseases;
3. Volunteers with informed consent.

Exclusion Criteria:

1. Patients combined with infection;
2. Patients with end-stage renal disease and undergoing renal replacement therapy
3. Patients with the history of thromboembolism;
4. Patients with malignant tumor and undergoing chemotherapy;
5. Patients with unmanageable hypertension (systolic pressure>200 mmHg or diastolic pressure>110mmHg);
6. Patients allergic to erythropoietin;
7. Patients injected erythropoietin within 2 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Study Chair — Nanjing First Hospital, Nanjing Medical University; Xin Wan, Doctor, Study Director — Nanjing First Hospital, Nanjing Medical University; Changchun Cao, Doctor, Study Director — Nanjing First Hospital, Nanjing Medical University; Xin Du, Doctor, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corwin HL, Gettinger A, Fabian TC, May A, Pearl RG, Heard S, An R, Bowers PJ, Burton P, Klausner MA, Corwin MJ; EPO Critical Care Trials Group. Efficacy and safety of epoetin alfa in critically ill patients. N Engl J Med. 2007 Sep 6;357(10):965-76. doi: 10.1056/NEJMoa071533. PMID 17804841
- [Background] de Seigneux S, Ponte B, Weiss L, Pugin J, Romand JA, Martin PY, Saudan P. Epoetin administrated after cardiac surgery: effects on renal function and inflammation in a randomized controlled study. BMC Nephrol. 2012 Oct 3;13:132. doi: 10.1186/1471-2369-13-132. PMID 23033926
- [Background] Drueke TB, Locatelli F, Clyne N, Eckardt KU, Macdougall IC, Tsakiris D, Burger HU, Scherhag A; CREATE Investigators. Normalization of hemoglobin level in patients with chronic kidney disease and anemia. N Engl J Med. 2006 Nov 16;355(20):2071-84. doi: 10.1056/NEJMoa062276. PMID 17108342
- [Background] Kaufman JS, Reda DJ, Fye CL, Goldfarb DS, Henderson WG, Kleinman JG, Vaamonde CA. Subcutaneous compared with intravenous epoetin in patients receiving hemodialysis. Department of Veterans Affairs Cooperative Study Group on Erythropoietin in Hemodialysis Patients. N Engl J Med. 1998 Aug 27;339(9):578-83. doi: 10.1056/NEJM199808273390902. PMID 9718376
- [Background] Kim JH, Shim JK, Song JW, Song Y, Kim HB, Kwak YL. Effect of erythropoietin on the incidence of acute kidney injury following complex valvular heart surgery: a double blind, randomized clinical trial of efficacy and safety. Crit Care. 2013 Oct 24;17(5):R254. doi: 10.1186/cc13081. PMID 24156702
- [Background] Oh SW, Chin HJ, Chae DW, Na KY. Erythropoietin improves long-term outcomes in patients with acute kidney injury after coronary artery bypass grafting. J Korean Med Sci. 2012 May;27(5):506-11. doi: 10.3346/jkms.2012.27.5.506. Epub 2012 Apr 25. PMID 22563215
- [Background] Togel FE, Ahlstrom JD, Yang Y, Hu Z, Zhang P, Westenfelder C. Carbamylated Erythropoietin Outperforms Erythropoietin in the Treatment of AKI-on-CKD and Other AKI Models. J Am Soc Nephrol. 2016 Nov;27(11):3394-3404. doi: 10.1681/ASN.2015091059. Epub 2016 Mar 16. PMID 26984884
- [Background] Song YR, Lee T, You SJ, Chin HJ, Chae DW, Lim C, Park KH, Han S, Kim JH, Na KY. Prevention of acute kidney injury by erythropoietin in patients undergoing coronary artery bypass grafting: a pilot study. Am J Nephrol. 2009;30(3):253-60. doi: 10.1159/000223229. Epub 2009 Jun 2. PMID 19494484
- [Background] Tasanarong A, Duangchana S, Sumransurp S, Homvises B, Satdhabudha O. Prophylaxis with erythropoietin versus placebo reduces acute kidney injury and neutrophil gelatinase-associated lipocalin in patients undergoing cardiac surgery: a randomized, double-blind controlled trial. BMC Nephrol. 2013 Jul 5;14:136. doi: 10.1186/1471-2369-14-136. PMID 23829828
- [Background] Tie HT, Luo MZ, Lin D, Zhang M, Wan JY, Wu QC. Erythropoietin administration for prevention of cardiac surgery-associated acute kidney injury: a meta-analysis of randomized controlled trials. Eur J Cardiothorac Surg. 2015 Jul;48(1):32-9. doi: 10.1093/ejcts/ezu378. Epub 2014 Oct 13. PMID 25312524

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Erythropoietin Group
Started | 51 | 50
Completed | 46 | 46
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Erythropoietin Group | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 18 | 18 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
serum creatinine [Mean (Standard Deviation); unit: μmo/L] | 74.5 (27.6) | 76.0 (26.2) | 75.2 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Kidney Injury
Description: Occurrence of acute kidney injury according to KDIGO guideline
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Control Group | Erythropoietin Group
Number analyzed (Participants) | 46 | 46
participants | 15 | 9

2. Secondary Outcome: Number of Participants With Renal Replacement Therapy
Description: suffering from severe acute kidney injury(3.0 times baseline OR Increase in serum creatinine to ≥4.0 mg/dl (≥353.6 mmol/l)), olignuria≥24 hours or anuria≥12 hours.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Control Group | Erythropoietin Group
Number analyzed (Participants) | 46 | 46
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: pulmonary infection, thrombotic events
Arm/Group | Control Group | Erythropoietin Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 10/46 | 9/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=46) | Erythropoietin Group (N=46)
Thrombotic events (Vascular disorders) | 0 (0) | 0 (0)
pulmonary infection (Infections and infestations) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03007537/Prot_SAP_000.pdf